CLINICAL TRIAL: NCT01900444
Title: Immunogenicity and Safety Exploration of a Booster Dose of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®) Given One Year After Primary Immunization in Healthy Children in South Korea
Brief Title: Study of a Booster Dose of IMOJEV® One Year After Primary Immunization in Healthy Children in South Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEC22; U1111-1127-7153 (Other: WHO)
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Japanese Encephalitis
Keywords: Japanese encephalitis; Japanese encephalitis chimeric virus vaccine; IMOJEV®
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IMOJEV Group (Experimental): Participants who received a single dose of IMOJEV in study JEC12 (NCT01396512) will receive a booster dose in this study.
  Interventions: Biological: IMOJEV

INTERVENTIONS:
Biological: IMOJEV — 0.5 mL, Subcutaneous
  Other Names: Japanese Encephalitis Chimeric Virus Vaccine

SUMMARY:
The aim of this study was to document the immunogenicity and safety of a booster dose of IMOJEV administered at least 12 months after the primary dose.

Primary objective:

* To describe the immune response to Japanese Encephalitis (JE) before and 28 days after a booster dose of IMOJEV administered at least 12 months after primary vaccination with IMOJEV.

Exploratory objectives:

* To describe the safety profile of a booster dose of IMOJEV® .

DETAILED DESCRIPTION:
Participants who previously participated in Study JEC12 (NCT01396512) and were primed with IMOJEV received a booster dose of IMOJEV at least 12 months after the primary dose. Participants were assessed for immune response before and on Day 28 after the booster dose and were monitored for safety through Day 28 post-vaccination for non-serious adverse events (AEs) and up to 6 months post-vaccination for serious AEs The duration of each participant's participation in the study was approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in study JEC12 and received 1 dose of IMOJEV at least 12 months before booster vaccination
* Age 2 to 4 years on the day of inclusion
* In good general health at the time of inclusion
* Informed Concent Form signed and dated by parent(s) or another legally acceptable representative(s)
* Subject and parent(s)/legally acceptable representative(s) able to attend all scheduled visits and comply with all study procedures.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical study investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the study vaccination
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Receipt of immune globulins, blood or blood-derived products in the past 3 months, that might interfere with the assessment of the immune response
* Previous vaccination against flavivirus disease, including JE, with another vaccine, except with IMOJEV® while participating in JEC12
* Administration of any anti-viral within 2 months preceding Visit 1 and up to the 4 weeks following the study vaccination
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination, except for inactivated influenza vaccination, which may be received at least 2 weeks before the study vaccine
* History of central nervous system disorder or disease, including seizures
* Planned receipt of any JE vaccine during the course of the study
* History of flavivirus infection (confirmed either clinically, serologically or virologically)
* Administration of systemic corticosteroids for more than 2 consecutive weeks within the 4 weeks preceding vaccination
* Thrombocytopenia, contraindicating vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating vaccination
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection 3 days before vaccination as well as the day of vaccination, according to Investigator judgment. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* In an emergency setting or hospitalized involuntarily
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2014-03-11 (Actual); Study Completion 2014-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur South Korea
Locations (8):
- South Korea (8):
  - Investigational Site 004, Gyeonggi-do
  - Investigational Site 010, Gyeonggi-do
  - Investigational Site 001, Seoul
  - Investigational Site 005, Seoul
  - Investigational Site 006, Seoul
  - Investigational Site 008, Seoul
  - Investigational Site 009, Seoul
  - Investigational Site 007, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 11 July 2013 to 27 September 2013 at 8 clinic centers in South Korea.
Pre-assignment Details: A total of 119 participants who met all inclusion and no exclusion criteria were enrolled and vaccinated.
Groups:
- Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®): Participants 2 to 4 years of age received one booster dose of IMOJEV® 1 year after primary immunization.
Period: Overall Study
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Started | 119
Completed | 116
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 119
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 2.62 (0.391)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 71
Region of Enrollment [Number; unit: Participants]
  South Korea | 119

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With JE Seroprotection Before and Following a Booster Dose of IMOJEV Given One Year After Primary Immunization
Description: JE virus neutralizing antibodies were measured using a 50% plaque reduction neutralization test (PRNT50). Seroprotection status for antibody levels against JE virus before and after IMOJEV vaccination was defined as antibody titers ≥ 10 (1/dilution).
Time Frame: Day 0 (pre-booster) and Day 28 post-booster injection
Population: Seroprotection rates were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Percentage of participants
  Pre-Booster | 93.5
  Post-Booster | 100.0

2. Primary Outcome: Percentage of Participants With JE Seroconversion Following a Booster Dose of IMOJEV Given One Year After Primary Immunization
Description: JE virus neutralizing antibodies were measured using PRNT50. Seroconversion was defined as a pre-vaccination titer <10 (1/dilution) and post-vaccination titer ≥10 (1/dilution, or pre-vaccination titer ≥10 (1/dilution) and a ≥4-fold increase of titers from pre- to post-vaccination.
Time Frame: Day 28 post-booster injection
Population: Seroconversion rates were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Percentage of participants | 94.6

3. Primary Outcome: Summary of Geometric Mean Titers of JE Virus Antibodies Following a Booster Dose of IMOJEV Given One Year After Primary Immunization
Description: JE virus neutralizing antibodies were measured using PRNT50 test.
Time Frame: Day 0 (pre-booster) and Day 28 post-booster injection
Population: Geometric mean titers of JE virus antibodies were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Titer
  Pre-Booster | 165 [116 to 235]
  Post-Booster | 8482 [6994 to 10286]

4. Primary Outcome: Summary of Geometric Mean Titer Ratios of JE Virus Antibodies Following a Booster Dose of IMOJEV Given One Year After Primary Immunization
Description: JE virus neutralizing antibodies were measured using PRNT50.
Time Frame: Day 0 (pre-booster) and Day 28 post-booster injection
Population: Geometric mean titer ratios of JE virus antibodies were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Ratio | 51.4 [37.3 to 71.0]

5. Primary Outcome: Percentage of Participants With JE Seroprotection Before and After a Booster Dose of IMOJEV Given At Different Intervals After Primary Immunization
Description: JE virus neutralizing antibodies were measured using PRNT50. Seroprotection was defined as neutralizing antibody titer ≥ 10 (1/dilution).
Time Frame: Day 0 (pre-booster) and Day 28 post-booster injection
Population: Seroprotection rates were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Percentage of participants
  Pre-Booster; ≥12 months and <18 months: number analyzed (Participants) | 53
  Pre-Booster; ≥12 months and <18 months | 92.5
  Post-Booster; ≥12 months and <18 months: number analyzed (Participants) | 53
  Post-Booster; ≥12 months and <18 months | 100.0
  Pre-Booster; ≥18 months and <24 months: number analyzed (Participants) | 38
  Pre-Booster; ≥18 months and <24 months | 94.7
  Post-Booster; ≥18 months and <24 months: number analyzed (Participants) | 38
  Post-Booster; ≥18 months and <24 months | 100.0
  Pre-Booster; ≥24 months: number analyzed (Participants) | 1
  Pre-Booster; ≥24 months | 100.0
  Post-Booster; ≥24 months: number analyzed (Participants) | 1
  Post-Booster; ≥24 months | 100.0

6. Primary Outcome: Percentage of Participants With JE Seroconversion Following a Booster Dose of IMOJEV Given At Different Intervals After Primary Immunization
Description: JE virus neutralizing antibodies were measured using PRNT50. Seroconversion was defined as a pre-vaccination titer <10 (1/dilution) and post-vaccination titer ≥10 (1/dilution, or pre-vaccination titer ≥10 (1/dilution) and a ≥4 fold increase from pre- to post-vaccination.
Time Frame: Day 28 post-booster injection
Population: Seroconversion rates were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Percentage of participants
  Post-Booster; ≥12 months and <18 months: number analyzed (Participants) | 53
  Post-Booster; ≥12 months and <18 months | 96.2
  Post-Booster; ≥18 months and <24 months: number analyzed (Participants) | 38
  Post-Booster; ≥18 months and <24 months | 92.1
  Post-Booster; ≥24 months: number analyzed (Participants) | 1
  Post-Booster; ≥24 months | 100.0

7. Primary Outcome: Summary of Geometric Mean Titers of JE Virus Antibodies Following a Booster Dose of IMOJEV At Different Intervals After Primary Immunization
Description: JE virus neutralizing antibodies were measured using PRNT50.
Time Frame: Day 0 (pre-booster) and Day 28 post-booster injection
Population: Geometric mean titers of JE virus antibodies were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Titer
  Pre-Booster; ≥12 months and <18 months: number analyzed (Participants) | 53
  Pre-Booster; ≥12 months and <18 months | 131 [5.00 to 5120]
  Post-Booster; ≥12 months and <18 months: number analyzed (Participants) | 53
  Post-Booster; ≥12 months and <18 months | 8199 [320 to 20480]
  Pre-Booster; ≥18 months and <24 months: number analyzed (Participants) | 38
  Pre-Booster; ≥18 months and <24 months | 239 [5.00 to 20480]
  Post-Booster; ≥18 months and <24 months: number analyzed (Participants) | 38
  Post-Booster; ≥18 months and <24 months | 8850 [160 to 20480]
  Pre-Booster; ≥24 months: number analyzed (Participants) | 1
  Pre-Booster; ≥24 months | 20.0 [20.0 to 20.0]
  Post-Booster; ≥24 months: number analyzed (Participants) | 1
  Post-Booster; ≥24 months | 10240 [10240 to 10240]

8. Primary Outcome: Summary of Geometric Mean Titer Ratios of JE Virus Antibodies Following a Booster Dose of IMOJEV Given At Different Intervals After Primary Immunization
Description: JE virus neutralizing antibodies were measured using PRNT50.
Time Frame: Day 0 (pre-booster) and Day 28 post-booster injection
Population: Geometric mean titer ratios of JE virus antibodies were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Number analyzed (Participants) | 92
Ratio
  Post-Booster; ≥12 months and <18 months: number analyzed (Participants) | 53
  Post-Booster; ≥12 months and <18 months | 62.3 [2.00 to 1024]
  Post-Booster; ≥18 months and <24 months: number analyzed (Participants) | 38
  Post-Booster; ≥18 months and <24 months | 37.0 [1.00 to 1024]
  Post-Booster; ≥24 months: number analyzed (Participants) | 1
  Post-Booster; ≥24 months | 512 [512 to 512]

ADVERSE EVENTS:
Time Frame: Solicited injection site reactions were collected from Day 0 to Day 7 and solicited systemic reactions from Day 0 to Day 14. Unsolicited AEs were collected from Day 0 to Day 28 for non-serious AEs and up to 6 months for serious AEs post-booster injection.
Description: The following pre-defined solicited adverse reactions were collected: Injection Site Pain, Erythema, and Swelling, as well as Fever, Headache, Malaise, and Myalgia. Solicited reactions are prelisted in the eCRF and considered to be related to vaccination, while unsolicited AsE are AEs that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or time to onset post-vaccination.
Arm/Group | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
All-Cause Mortality (participants affected / at risk) | 0/119
Serious Adverse Events (participants affected / at risk) | 4/119
Other Adverse Events (participants affected / at risk) | 48/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®) (N=119)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Henoch Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®) (N=119)
Nasopharyngitis (Infections and infestations) | 33 (36)
Injection site Pain (General disorders) | 34 (34)
Injection site Erythema (General disorders) | 17 (17)
Injection site Swelling (General disorders) | 10 (10)
Fever (General disorders) | 15 (15)
Headache (Nervous system disorders) | 22 (22)
Malaise (General disorders) | 48 (48)
Myalgia (General disorders) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications